CLINICAL TRIAL: NCT04503317
Title: Influence of Exercise Training Combined With Laser Phototherapy on Coagulation Profile in Senior Individuals With Obesity: A Randomized Clinical Trial
Brief Title: Effect of Phototherapy With Exercise on Coagulation in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/002724
Record Dates: First submitted 2020-07-26; First posted 2020-08-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Hypercoagulability; Obesity
MeSH Terms: conditions — Thrombophilia; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active acupuncture low level laser and aerobic exercise (Experimental): active acupuncture, low level laser and aerobic exercise
  Interventions: Device: active acupuncture low level laser in addition to nasal laser irradiation; Other: treadmill exercise
- aerobic exercise (Active Comparator): aerobic exercise
  Interventions: Other: treadmill exercise

INTERVENTIONS:
Device: active acupuncture low level laser in addition to nasal laser irradiation — laser consists of a semiconductor and operates at a wavelength of 650 nanometre. The laser installed in the watch comprises 10 individual laser beams for the wrist and an additional adapter for nasal stimulation. The output power is 5 megawatt, but it can also be adjusted. The device operates at an ambient temperature of -20 to +40 ° C and relative humidity of ≤ 85%. The laser watch can be used for a variable irradiation period of 10-60 min. applied on specific acupuncture points ( acupuncture point, Radial artery acupuncture points, and ulnar artery acupuncture points) combined with nasal laser irradiation at the same time with treadmill aerobic exercise, once per day, 3 times per week for three months
  Arms: active acupuncture low level laser and aerobic exercise
Other: treadmill exercise — aerobic exercise once per day, 3 times per week for three months

SUMMARY:
It is an interventional study in which 60 obese elderly patients (30 male & 30 female) estimated to enroll according to random allocation and divided into two groups. The study group will receive active acupuncture low level laser in addition to nasal laser irradiation and aerobic exercises while the control group will aerobic exercises. The laser consists of a semiconductor and operates at a wavelength of 650 nanometre. The laser installed in the watch comprises 10 individual laser beams for the wrist and an additional adapter for nasal stimulation. The output power is 5 megawatt, but it can also be adjusted. The device operates at an ambient temperature of -20 to +40 ° C and a relative humidity of ≤ 85%. The laser watch can be used for a variable irradiation period of 10-60 min. the device will be applied on specific acupuncture points ( acupuncture point, Radial artery acupuncture points, and ulnar artery acupuncture points) combined with nasal laser irradiation at the same time, once per day, 3 times per week for three months

DETAILED DESCRIPTION:
PURPOSE:

To determine whether low level laser light therapy is effective as an adjunctive therapy on countering hypercoagulable state parameters (fibrinogen, bleeding time, Prothrombin time) and total cholesterol (, d-dimer and c-reactive protein) as preventive strategy of venous thromboembolism incidence in obese elderly patients

BACKGROUND:

In the general population the annual incidence of venous thrombosis (VT) approximates 1 in 1000 persons and appears to be increasing over time. Notably, incidence rates rise exponentially with age with an approximate 7- to 10-fold increase from less than 55 years to greater than 75 years. Aging is associated with increased levels of coagulation factors and decrease in natural anticoagulant factors. This strongly supports that age-related hypercoagulable state occurs in elderly.

Blood coagulation plays a critical role not only in homeostasis but also in many physiological and pathological conditions. Blood coagulation potential in humans reaches a young adult level around the time of weaning, followed by a gradual increase during young adulthood and an almost 2-fold increase by old age.

Fibrinogen may contribute to the cardiovascular risk due to their influence on blood viscosity, platelet aggregation, low-density lipoprotein deposition, blood vessel diameter and cell proliferation. Most of the factors that cause venous thromboembolism are related to changes in blood flow and changes in the composition of the blood.

In recent years, an innovative technology using low-level laser light has garnered an exceptional level of interest across myriad medical disciplines because of its unique ability to modulate cellular metabolism, therefore inducing beneficial clinical effects

Low level laser radiation has particular effect on blood viscosity by changing the sizes of erythrocyte aggregates which lead to an increase in the blood flow velocity in the human body. There are several reasons for the increase in the blood microcirculation under irradiation. One of the major reasons is the activation of the respiratory chains of cells leading to a cascade of biochemical reactions that resulting in an increase in the permeability of erythrocyte membranes and an increase in the concentration of oxygen in the bio tissues.

HYPOTHESES:

countering hypercoagulable state parameters (fibrinogen, bleeding time, Prothrombin time) and total cholesterol (, d-dimer and c-reactive protein) as a preventive strategy of venous thromboembolism incidence in obese elderly patients

RESEARCH QUESTION:

Does low level laser therapy with aerobic exercises influence on obese elderly patients' hemostatic state parameters as coagulation profile ((fibrinogen, bleeding time, Prothrombin time) and total cholesterol (, d-dimer and c-reactive protein) as prevention of venous thromboembolism in the obese elderly patient

ELIGIBILITY:
Inclusion Criteria:

* • aged from 60 to 75 y

  * • sedentary individuals
  * Body mass index 30-39.9 kg/m2

Exclusion Criteria:

* • The exclusion criteria were as follows: smokers, diabetes, drinking alcohol, presence of uncontrolled hypertension or cardiovascular diseases, weight loss program participation for at least 6 months prior to the current study, medications affecting blood coagulation or body weight, recent or chronic active disease, cognitive impairment, presence of malignant disease, blood donation, or participation in any other research during the previous 90 days of the current study Individuals suffering from hepatic, renal, cardiac, chest, and endocrine diseases, as well as musculoskeletal disease

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
fibrinogen | 12 weeks
  measuring by blood analysis change of fibrinogen
Prothrombin time and partial thromboplastin time | 12 weeks
  change of Prothrombin time and partial thromboplastin time by blood analysis
total cholesterol | 12 weeks
  change of total cholesterol by blood analysis
d-dimer | 12 weeks
  change of d-dimer by blood analysis
c-reactive protein | 12 weeks
  change of c-reactive protein by blood analysis

SECONDARY OUTCOMES:
body mass index | 12 weeks
  measuring the participants' weights (in kilogram) and heights (in meter)
Waist-Hip ratio | 12 weeks
  It is measured by dividing the participants' circumferences of their waists and hips

CONTACTS AND LOCATIONS:
Overall Officials: marwa m elsayed, phd, Principal Investigator — physical therapy faculty Cairo university
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: after completing the study by one year
Access Criteria: journal published the study
URL: http://Scholar.cu.edu.eg/p_t

REFERENCES:
- [Derived] Elsayed MM, Abdallah GA, Hassan SS, Nagy EN. Effect of exercise training with laser phototherapy on homeostasis balance resistant to hypercoagulability in seniors with obesity: a randomized trial. Sci Rep. 2023 Mar 3;13(1):3592. doi: 10.1038/s41598-023-30550-x. PMID 36869148